CLINICAL TRIAL: NCT02574325
Title: A Study to Assess ARI-3037MO on Hepatic Fat Metabolism in Patients With Dysglycemia and Evidence of Hepatic Steatosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Arisaph Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ARI-3037MO-006
Record Dates: First submitted 2015-10-08; First posted 2015-10-12 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2015-10

CONDITIONS: Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- ARI-3037MO (Experimental): ARI-3037MO
  Interventions: Drug: ARI-3037MO

INTERVENTIONS:
Drug: Placebo — Control
  Arms: Placebo
Drug: ARI-3037MO — Treatment
  Arms: ARI-3037MO

SUMMARY:
Primary objective To investigate the effect of a 24-week, twice daily dosing regimen of ARI-3037MO compared to placebo on plasma triglyceride (TG) levels, liver enzymes and hepatic fat content in patients with dysglycemia and hepatic steatosis due to nonalcoholic fatty liver disease (NAFLD) or nonalcoholic steatohepatitis (NASH). Secondary Objective To investigate the safety and tolerability of a 24-week, twice daily dosing regimen of ARI-3037MO compared to placebo in patients with dysglycemia and evidence of NAFLD or NASH.

DETAILED DESCRIPTION:
This randomized,double-blind, placebo-controlled study will enroll 36 men and women with a diagnosis of NAFLD orNASH. The study will be conducted over a period of approximately 28 wks and will include:a Screening Phase (Days -14to -1); a 24-week long Treatment Phase, during which patients will be randomly assigned to receive ARI-3037MO or placebo; an End-of-study Visit (ESV) scheduled 2 wks after the end of the Treatment Phase The Screening Phase will include 2 visits. Visit 1:There will be an initial assessment of a patient's eligibility for participation in the study. A complete medical history will be obtained and prospective study patients will undergo physical examinations and laboratory evaluations. For patients who have had a liver biopsy in the 6months prior to Visit 1, the histology findings, i.e., NAS, steatosis score and fibrosis score will be recorded. Visit 2:Approximately 1 week after Visit 1, and after the results of clinical laboratory screening test results have been reviewed by the Principal Investigator (PI), patients will be contacted to advise them of their eligibility to continue in the study. Eligible patients will undergo liver magnetic resonance imaging (MRI) to assess intrahepatic fat content. Treatment Phase Patients with MRI results showing intrahepatic fat content of ≥10% will be entered into the Treatment Phase of the study. The Treatment Phase will include 4 outpatient visits over a period of 24 weeks. Visit 3:Patients will be randomly assigned to receive ARI-3037MO or placebo on Day 1 of a 24-week long outpatient treatment period. Baseline assessments, including FibroTest®, FibroScan® and clinical laboratory tests, will be performed, and patients will take study drug twice daily. Visits 4, 5 and 6: During the Treatment Phase, patients will visit the study clinic at 4, 12 and 24 weeks (± 4 days) after Day 1 for evaluations and examinations and to collect study drug. Twenty-four weeks after the start of dosing, at the end of the Treatment Phase, patients will undergo a follow-up MRI and FibroScan† to assess change from baseline in intrahepatic fat content and liver fibrosis, respectively.

†If FibroScan equipment is available at the study site End-of-Study Visit Visit 7:An ESV will occur 2 weeks (± 4 days) after the end of the Treatment Phase.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients ≥ 18 years of age at study entry
2. Female patients must be of nonchildbearing potential
3. Have a stable diet and agree to maintain this diet throughout the study
4. Have not gained or lost ≥ 10 lbs (4.5 kg) of body weight within 6months prior to Screening Visit 1
5. Have a body mass index (BMI) between 28 and 45 kg.m-2, inclusive
6. Have elevated alanine aminotransferase (ALT) levels. For men: 50 IU/L to 250 IU/L, inclusive. For women: 40 IU/L to 240 IU/L, inclusive.
7. Have HbA1c of < 9.5
8. Have a intrahepatic fat content of ≥ 10% confirmed by liver MRI
9. If taking antidiabetic therapies (excluding thiazolidines as per exclusion Criterion No. 13), i.e., metformin, sulfonylureas, dipeptidyl peptidase-4 inhibitors, insulin; must be on a stable dose for at least 3months prior to Screening Visit 1. Similarly, if taking lipid lowering therapies; must be on a stable dose for at least 3 months prior to Screening Visit 1.
10. Understands the study requirements and the treatment procedures, is willing to comply with all protocol-required evaluations and provides written informed consent before any study specific tests or procedures are performed

Exclusion Criteria:

1. A history of hepatic disease such as chronic hepatitis C virus or concurrent active hepatitis B virus (i.e., serum positive for hepatitis B surface antigen)
2. Autoimmune hepatitis
3. Primary biliary cirrhosis
4. Sclerosing cholangitis
5. Hereditary hemochromatosis
6. History of chronic / repeat blood transfusion (i.e., ≥ 20 units of blood)
7. Alpha-1 anti-trypsin deficiency
8. Wilson's disease
9. Thyroid disease
10. Bariatric surgery within 5 years prior to Screening Visit 1
11. Hepatic disease due to substance abuse
12. Have any concurrent disease or condition not listed above that, in the opinion of the PI, would make the patient unsuitable for participation in the study
13. Currently taking thiazolidines (glitazone therapy, i.e., Rosiglitazone, Pioglitazone)
14. Liver biopsy in the past 90 days with negative results for cirrhosis and steatosis
15. No evidence of hepatic decompensation or elevated serum bilirubin > 1.5 times the upper limit of normal
16. Estimated glomerular filtration rate < 60 mL/min according to the Modification of Diet in Renal Disease equation
17. Known substance abuse
18. Current smoker or a history of smoking (> 10 cigarettes, > 3 cigars or > 3 pipes/day)
19. Current consumption of > 3 units of alcohol per day (> 21 units per week) for men and > 2 units of alcohol per day (> 14 units per week) for women
20. Currently participating in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy as measured by change in intra hepatic fat content | 24 wks
  Change in intra hepatic fat content by MRI
Efficacy as measured by change in plasma ALT levels | 24 wks
  Change in plasma ALT levels from baseline
Efficacy as measured by change in plasma TG levels | 24 wks
  Change in plasma TG levels from baseline

SECONDARY OUTCOMES:
Safety as measured by the occurrence of flushing (number of episodes) and itching (number of episodes) | 24 wks
  Occurrence of cutaneous symptoms
Safety as measured by effect of ARI-3037MO on on glycemic control | 24 wks
  Change in HbA1c levels from baseline
Safety as measured by effect of ARI-3037MO on serum bilirubin, alkaline phosphatase, Prothrombin time and plasma albumin levels | 24 wks
  Change of liver function tests from baseline
Safety as measured by effect of ARI-3037MO on gastrointestinal systems; episodes of nausea, vomiting and diarrhea | 24 wks
  occurrence of GI symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Gastroenterology & Hepatology CRU, St Louis University, St Louis, Missouri, United States